CLINICAL TRIAL: NCT07131943
Title: Comparison Between Radiofrequency and Ultrasound on Shoulder Pain, Range of Motion, and Functional Outcomes in Patients With Stroke
Brief Title: Radiofrequency vs. Ultrasound Therapy for Shoulder Joint in Stroke Patients: A Comparative Clinical Trial
Acronym: TECAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Rewan Magdy Aloush, Demonestrator for Physical Therapy for Neurology and Its Surgery, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RADIOFREQUENCY AND ULTRASOUND
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Stroke ( 3 Months After Onset); Stroke in Patients: New Tool to Evaluate the Impact in Their Life
Keywords: Stroke; Hemiplegia; TECAR; Radiofrequency; Shoulder Pain
MeSH Terms: conditions — Stroke; Hemiplegia; Shoulder Pain | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Fourty-five hemiplegic patients with shoulder pain post- stroke from both sexes will participate in this study.
  * The patients will be older than 18 years old (30-60 years old)
  * The presence of sub-acute shoulder pain (more than 3 months).
  * Sub-acute stroke survivors (3 months post-stroke).
  * score of 1|1+ points on the Modified Ashworth Scale (MAS) on shoulder joint.
  * Stage 2 or above according to Brunnstrom function assessment of shoulder joint
  * All conducted patients experienced a single stroke during the last 3 months with cognitive capacity that will enable them to comprehend and follow the instructions (Mini-Mental Scale score > 24).
  Therapeutic Equipment and tools TECAR (Transfer Electrical Capacitive and Resistive) therapy and ultrasound therapy are advanced non-invasive therapeutic modalities used in physiotherapy to accelerate tissue healing and pain relief. TECAR therapy utilizes radiofrequency energy to generate deep endogenous heat, enhancing blood flow.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (GI)= 15 will be treated by Radiofrequency TECAR Therapy (Experimental): Group (GI) will be treated by Radiofrequency TECAR Therapy on shoulder joint as well as Designed Physical Therapy Program
  Interventions: Device: Radiofrequency
- Group (GII)= 15 will be treated by Ultrasound Therapy (Experimental): Group (GII) will be treated by Ultrasound Therapy on shoulder joint as well as Designed Physical Therapy Program
  Interventions: Device: Ultrasound
- Group (GIII)= 15 will be treated by Designed Physical Therapy Program, (Experimental): Group (GIII) will be treated by Designed Physical Therapy Program, all outcomes' measures will be assessed pre and post treatment.
  Interventions: Other: The designed physical therapy program

INTERVENTIONS:
Device: Radiofrequency — Radiofrequency (TECAR) therapy is a non-invasive, non-ablative treatment that uses electromagnetic energy to generate endogenous heat, promoting increased blood flow and tissue healing in both superficial and deep tissues. With a long wavelength and low frequency (300 KHz to 1 MHz), it can penetrate deeply into muscles, tendons, and bones, making it suitable even in acute conditions. TECAR operates in two modes: capacitive (targeting soft tissues rich in electrolytes) and resistive (targeting high-resistance tissues like bones and tendons). The therapy stimulates natural repair processes by inducing ion flow and micro-hyperemia, leading to the release of endorphins and cortisone, which help reduce pain, inflammation, and edema, while enhancing immune response and tissue regeneration.
  Arms: Group (GI)= 15 will be treated by Radiofrequency TECAR Therapy
Device: Ultrasound — The ultrasound waves accelerate healing, increasing local vascularity and improving several other characteristics, including energy absorption capacity and maximum rupture resistance tension, increased collagen synthesis, fibroblast proliferation, release of growth factors stimulated by mast cell degranulation and improved response of platelets and macrophages anticipating the proliferative and remodeling phase. 1-MHz continuous ultrasound, with a half-value depth of approximately 2.3 cm, is frequently used to treat deep tissues that are approximately 2.3 to 5 cm deep.
  Other Names: US
  Arms: Group (GII)= 15 will be treated by Ultrasound Therapy
Other: The designed physical therapy program — The designed physical therapy program focuses on improving upper limb mobility and stability through a structured set of exercises targeting the shoulder joint. It includes prolonged stretching performed in a seated position to extend the thumb, fingers, wrist, elbow, and shoulder, along with scapular mobilization in side-lying and stretching of internal rotators in a supine position. The stretching progression begins with external rotation at 45° abduction and advances to 90° abduction and full reach toward the ground if pain-free. Joint stabilization exercises involve resistance band movements in various shoulder and elbow positions, including controlled abduction, flexion, scapular movements, and external rotation, all aimed at enhancing joint control and muscular coordination.
  Other Names: Treatment Exercises
  Arms: Group (GIII)= 15 will be treated by Designed Physical Therapy Program,

SUMMARY:
The purpose of the current study is to:

Compare between radiofrequency (TECAR) therapy and ultrasound on Shoulder Pain, Range of Motion and Functional Outcome in Patients with stroke.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death worldwide and a major contributor to long-term disability, particularly affecting upper limb function in about 70% of survivors. Among post-stroke complications, hemiplegic shoulder pain (HSP) is notably challenging, affecting 30-65% of patients and often resulting from structural injuries, poor posture, or conditions like rotator cuff impingement and shoulder-hand syndrome. HSP is linked to reduced arm function, depression, and diminished quality of life. Therapeutic approaches such as TECAR therapy and therapeutic ultrasound aim to alleviate pain and promote tissue healing through deep heat and mechanical effects. Assessment tools like the algometer, Numerical Rating Scale (NRS), digital goniometer, and the Shoulder Pain and Disability Index (SPADI)-including its validated Arabic version-are reliable methods for evaluating pain, joint mobility, and functional disability in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Fourty-five hemiplegic patients with shoulder pain post- stroke from both sexes will participate in this study.
* The patients will be older than 18 years old (30-60 years old)
* The presence of sub-acute shoulder pain (more than 3 months).
* Sub-acute stroke survivors (3 months post-stroke).
* score of 1|1+ points on the Modified Ashworth Scale (MAS) on shoulder joint.
* Stage 2 or above according to Brunnstrom function assessment of shoulder joint
* All conducted patients experienced a single stroke during the last 3 months with cognitive capacity that will enable them to comprehend and follow the instructions (Mini-Mental Scale score > 24).

Exclusion Criteria:

* The following patients will be excluded from the study patients with:

  * Bilateral adhesive capsulitis
  * Systemic diseases such as rheumatoid arthritis, malignancies, heart diseases, infections, coagulation disorders, full rotator cuff tears
  * A history of recent shoulder surgery, neurological problems involving the upper extremity, shoulder joint osteoarthritis
  * Upper extremity fractures, cervical radiculopathy
  * Impaired sensation, having a heart pacemaker, pregnancy
  * Injuries in the upper limbs
  * Other neurological diseases or cancer
  * Osteosynthesis material or pacemaker
  * Botulinum toxin or antispastic treatment 3 months prior to studying.
  * Any contraindication to massage and Tecar as skin infections, inflammatory vascular diseases, or acute inflammation.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
Digital Goniometer for shoulder range of motion | 4 Weeks
  The digital goniometer (Baseline 12-1027 USA) will be used to assess range of motion (ROM) of the shoulder joint. The device consists of fixed arm, movable arm and screen. The device converts the angular displacement of the joint (represented in the degree of change of the angle between the two arms of the device) into an electric signal readout which is produced in a simple digital form.
  The device is the most accurate and objective method of ROM measurement with excellent inter-rater and intra-rater ranged from 0.89 to 0.98
The pressure algometer | 4 weeks
  The pressure algometer, specifically the hand-held Baseline® model, is a reliable and valid tool used to objectively measure pressure pain thresholds (PPT). It features a pistol-style grip and a pressure-sensitive gauge with a 0.785 cm² rubber tip. The device applies gradual, consistent manual force to determine the minimal pressure at which a sensation of pressure turns into pain. This method is widely used in clinical settings due to its strong correlation with pain intensity and excellent inter-rater reliability, making it a dependable tool for assessing pain sensitivity.
Numerical Rating Scale (NRS): | 4 weeks
  Numerical Rating Scale (NRS):
  For pain Threshold will be assessed by Numeric pain rating scale (NPRS) is an 11-point (0-10) Scale will be used to measure pain. Patients verbally will select value between (0-10) based on intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline
Functional Outcome and disability / Shoulder pain and Disability Index (SPADI) | 4 weeks
  The Shoulder Pain and Disability Index (SPADI) is a 13-item questionnaire used to assess the intensity of shoulder pain and the degree of functional disability. It includes two subscales: five questions evaluating pain severity and eight questions assessing difficulty with daily activities involving upper limb use. Patients mark their responses on a 10 cm visual analogue scale, with scores ranging up to 50 for pain, 80 for disability, and a total of 130, all expressed as percentages. SPADI has demonstrated strong validity and reliability, including in its Arabic version, with an intra-rater reliability coefficient of 0.89, making it a dependable tool for clinical and research use.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Delta University, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: No